CLINICAL TRIAL: NCT06196489
Title: Nicotine Cessation: Adapting a Counseling Program for Emerging Adults
Brief Title: Adapting an Intervention for Vaping in Young Veterans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: University of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VeteransMRF; T31P1525 (Other Grant/Funding Number: University of California)
Record Dates: First submitted 2023-12-13; First posted 2024-01-09 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: E Cigarette Use
Keywords: Veteran; e-cigarette; vaping; young adult
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telephone (Experimental): Participants assigned to this group will receive the adapted intervention by telephone.
  Interventions: Behavioral: adapted vaping cessation intervention
- Video (Experimental): Participants assigned to this group will receive the adapted intervention by video telehealth.
  Interventions: Behavioral: adapted vaping cessation intervention

INTERVENTIONS:
Behavioral: adapted vaping cessation intervention — Behavioral intervention for vaping cessation

SUMMARY:
The objective of this proposal is to adapt an evidence-based combustible tobacco counseling intervention following an evidence-based process to include e-cigarette use and update its components for emerging adults (EA).

1. Examine factors related to e-cigarette use, barriers to cessation, and facilitators of use of cessation services among an EA population.
2. Beta-test an initial version of the intervention, delivered via video telehealth and telephone, to examine usability and acceptability.

DETAILED DESCRIPTION:
Use of electronic nicotine products (ENDS) has increased dramatically especially among young adults (EA- aged 18-30) and has been found to lead to immediate harmful health effects and increased addiction to combustible cigarette use. To date no research-tested interventions have been developed for helping people stop use of electronic nicotine products. Emerging adulthood is a developmental period that can lead to adoption of health risk behaviors.

This proposal aims to address nicotine addiction by adapting an evidence-based counseling cessation intervention developed by the American Cancer Society (ACS) for a general population of combustible tobacco smokers, but found to be effective in EA. We will test two methods of providing counseling to participants: video telehealth or telephone. Primary outcome: Compared to self-help guide only, at 3 month follow-up, we hypothesize that participants in either counseling arm will have higher rates as compared to self-help only control of 7-day abstinence from using any nicotine product.

This study fills a critical gap in ENDS research and will provide a model for further research into all-nicotine cessation in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* daily e-cigarette user for at least the past 6 months
* 18-30 years old
* willing to enroll in a program to quit nicotine use within 30 days
* owns smartphone or computer/tablet with camera and internet connectivity
* English speaker

Exclusion Criteria:

* ICD-10 diagnosis of dementia
* current use of combustible tobacco products at least weekly

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
e-cigarette use frequency | end of treatment (8 weeks post-baseline) and 30 days thereafter
  number of days using e-cigarettes in the past 7 days at the time of assessment
e-cigarette use quantity | end of treatment (8 weeks post-baseline) and 30 days thereafter
  number of e-cigarette uses per day
Client Satisfaction Questionnaire (CSQ-8) | end of treatment (8 weeks post-baseline) and 30 days thereafter
  Participant satisfaction ratings; higher scores indicate greater satisfaction with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Neal M Doran, PhD, Principal Investigator — Veterans Medical Research Foundation
Locations (1):
- Veterans Medical Research Foundation, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Sample size is sufficiently small that sharing could threaten confidentiality.

REFERENCES:
- [Background] Palmer AM, Tomko RL, Squeglia LM, Gray KM, Carpenter MJ, Smith TT, Dahne J, Toll BA, McClure EA. A pilot feasibility study of a behavioral intervention for nicotine vaping cessation among young adults delivered via telehealth. Drug Alcohol Depend. 2022 Mar 1;232:109311. doi: 10.1016/j.drugalcdep.2022.109311. Epub 2022 Jan 19. PMID 35123362
- [Background] Kinouani S, Leflot C, Vanderkam P, Auriacombe M, Langlois E, Tzourio C. Motivations for using electronic cigarettes in young adults: A systematic review. Subst Abus. 2020;41(3):315-322. doi: 10.1080/08897077.2019.1671937. Epub 2019 Oct 22. PMID 31638872
- [Background] Harrell PT, Brandon TH, Stark SE, Simmons VN, Barnett TE, Quinn GP, Chun S. Measuring vaping-related expectancies in young adults: Psychometric evaluation of the Electronic Nicotine Vaping Outcomes (ENVO) scale. Drug Alcohol Depend. 2023 May 1;246:109861. doi: 10.1016/j.drugalcdep.2023.109861. Epub 2023 Mar 29. PMID 37028105
- [Background] Cuccia AF, Patel M, Amato MS, Stephens DK, Yoon SN, Vallone DM. Quitting e-cigarettes: Quit attempts and quit intentions among youth and young adults. Prev Med Rep. 2021 Jan 5;21:101287. doi: 10.1016/j.pmedr.2020.101287. eCollection 2021 Mar. PMID 33489721
- [Background] Buu A, Hu YH, Wong SW, Lin HC. Comparing American college and noncollege young adults on e-cigarette use patterns including polysubstance use and reasons for using e-cigarettes. J Am Coll Health. 2020 Aug-Sep;68(6):610-616. doi: 10.1080/07448481.2019.1583662. Epub 2019 Mar 25. PMID 30908151
- [Background] Bandi P, Star J, Minihan AK, Patel M, Nargis N, Jemal A. Changes in E-Cigarette Use Among U.S. Adults, 2019-2021. Am J Prev Med. 2023 Aug;65(2):322-326. doi: 10.1016/j.amepre.2023.02.026. Epub 2023 Apr 18. PMID 37479423